CLINICAL TRIAL: NCT01883700
Title: Variability of Acute Response to Equicaloric Test Meals Varying in Glycemic Index and Glycemic Load on Postprandial Glycemia, Arterial Stiffness and Blood Pressure in Healthy Adults
Brief Title: Acute Vascular Response To Meals Varying In Glycemic Index And Glycemic Load
Acronym: HILO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 10-028
Record Dates: First submitted 2013-02-22; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Healthy; Glycemic Index; Glycemic Load; Blood Glucose; Arterial Stiffness
MeSH Terms: interventions — Oils; Egg White

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low-GI, High-GL Meal (Experimental): Boiled Pasta
  Interventions: Other: Boiled Pasta
- Low-GI, High GL Meal (Experimental): Boiled Chickpeas with Oil
  Interventions: Other: Boiled Chickpeas with Oil
- High-GI, High-GL Meal (Experimental): Instant Mashed Potatoes
  Interventions: Other: Instant Mashed Potatoes
- High-GI, Low-GL Meal (Experimental): Instant Mashed Potatoes with Egg Whites
  Interventions: Other: Instant Mashed Potatoes with Egg Whites

INTERVENTIONS:
Other: Boiled Pasta
  Other Names: Italpasta Fusilli
  Arms: Low-GI, High-GL Meal
Other: Boiled Chickpeas with Oil
  Other Names: Irresistibles Life Smart Chick Peas
  Arms: Low-GI, High GL Meal
Other: Instant Mashed Potatoes
  Other Names: Betty Crocker Mashed Potatoes Homestyle
  Arms: High-GI, High-GL Meal
Other: Instant Mashed Potatoes with Egg Whites
  Other Names: Betty Crocker Mashed Potatoes Homestyle; Naturegg Simply Egg Whites 100% Pure Liquid Egg Whites
  Arms: High-GI, Low-GL Meal

SUMMARY:
This study examines the effects of carbohydrate type (high- or low-Glycemic Index (GI)) and amount (high- or low-Glycemic Load (GL)) have on blood glucose levels, blood pressure and arterial stiffness in healthy individuals. It will also determine whether subjective ratings such as test meal palatability and hunger are related to changes in blood glucose. The investigators hypothesize that: (1) High-GI meals, regardless of GL, will increase arterial stiffness; low-GI meals, regardless of GL, will have a neutral or lowering effect on arterial stiffness (augmentation index). (2) High-GI meals, regardless of GL, will have an elevating effect on both central and peripheral blood pressures. (3) The incremental area under the curve for blood glucose will show most significant differences between high-GI, high-GL and low-GI, low-GL meals at 30 and 90 min.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age 18 - 75 years
* BMI 18 - 25 kg/m2
* brachial systolic blood pressure < 140 mmHg
* brachial diastolic blood pressure < 90 mmHg

Exclusion Criteria:

* primary hypertension
* diabetes
* allergy or sensitivity to any foods to be used in the study
* gastrointestinal disorders
* chronic kidney disease
* liver disease
* hepatitis
* estrogen-sensitive cancer
* heavy alcohol use
* sleep apnea
* bleeding disorders
* planned surgery (within time frame of study)
* angina
* Congestive Heart Failure
* coronary revascularization
* peripheral vascular disease and/or coronary/cerebrovascular events within the previous 6 months
* positive HIV diagnosis
* prescription of anti-depressants, anti-hypertensives, anti-coagulant medications, diuretics, sympathomimetics, herbal therapies, vitamin or K supplementation, medication affecting NO synthesis
* chronic use or prescription of NSAIDs
* women of childbearing potential must not be pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
To measure postprandial changes in augmentation index (AIx) to determine the acute effect of high- and low-GI and high- and low-GL meals on arterial stiffness. | 4 separate mornings, measurements taken at baseline and at 60, 120, 180 and 240 minutes

SECONDARY OUTCOMES:
To determine the acute effect of high- and low-GI and high- and low- GL meals on central and peripheral blood pressure | 4 separate mornings, measurements taken at baseline, 60, 120, 180 and 240 minutes.

OTHER OUTCOMES:
To determine whether the effects of high- and low-GI and high- and low-GL meals on postprandial glycemia are correlation with arterial stiffness, central and peripheral blood pressure. | 4 separate mornings, measurements taken at baseline 15, 30, 45, 60, 90, 120, 180 and 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Jenkins, PhD, RD, Principal Investigator — Unity Health Toronto; Vladimir Vuksan (Co-Investigator), PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada